CLINICAL TRIAL: NCT00207142
Title: A Phase IV, Open-Label, Randomized, Multicenter Trial Assessing the Efficacy of a Treatment Maintenance Phase With Unboosted vs. Boosted Reyataz After an Induction Phase With Reyataz and Ritonavir in Treatment Naive HIV Patients (the INDUMA Study)
Brief Title: Induction-Maintenance With Atazanavir in HIV Naïve Patients (The INDUMA Study)
Acronym: INDUMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-136
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: Treatment Naive; HIV-1 infected treatment naive patients
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Switch (Active Comparator): ATV 400 mg + 2 NRTIs (TBD), ATV once daily, NRTIs (TBD)
  Interventions: Drug: Atazanavir + 2 NRTIs
- Continuation (Active Comparator): ATV 300 mg + RTV 100 mg + 2 NRTIs (TBD), ATV and RTV once daily, NRTIs (TBD)
  Interventions: Drug: Atazanavir + Ritonavir + 2 NRTIs
- Rescue (Other): ATV 300 mg + RTV 100 mg + 2 NRTIs (TBD), ATV and RTV once daily, NRTIs (TBD)
  Interventions: Drug: Atazanavir + Ritonavir + 2 NRTIs

INTERVENTIONS:
Drug: Atazanavir + 2 NRTIs — Capsules, tablets, Oral, 48 weeks (after a 26-to-30-week induction phase with ATV 300 mg + RTV 100 mg + 2 NRTIs)
  Other Names: Reyataz
  Arms: Switch
Drug: Atazanavir + Ritonavir + 2 NRTIs — Capsules, tablets, Oral, 48 weeks (after a 26-to-30-week induction phase with ATV 300 mg + RTV 100 mg + 2 NRTIs)
  Other Names: Reyataz
  Arms: Continuation; Rescue

SUMMARY:
The purpose of this study is to compare the proportion of subjects with HIV-1 RNA viral load < 50 c/mL through Week 48 of the Maintenance Phase among HIV-infected subjects with an initial undetectable viral load following an Induction Phase with an ATV/RTV containing HAART regimen, when switched to ATV versus remaining on ATV/RTV, whilst continuing their previous NRTI backbone.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive HIV-1 infected subjects ( < 10 days of treatment with any ARV).
* Subjects who have an HIV-1 RNA level ≥ 5000 c/mL at screening.
* Subjects who have a CD4 count ≥ 50 cells/mm3.
* Men and women, ages 18 years of age or older (or minimum age as determined by local regulatory or as legal requirements dictate).
* Both females of child-bearing potential and males must utilize effective barrier contraception. Other contraception in addition to barrier methods is permitted; refer to the Investigator Brochure for details regarding potential interactions with ATV and some oral contraceptives

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study.
* WOCBP using a prohibited contraceptive method. Caution is warranted with coadministration of oral contraceptives (ethinyl estradiol and norethindrone) - see Investigator Brochure for details
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment
* Primary HIV infection
* Medical History and Concurrent Diseases
* Active alcohol or substance use sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis Physical and Laboratory Test Findings
* Screening laboratory values measured as follows:
* Grade IV glucose,
* Grade IV electrolytes,
* Grade IV transaminases,
* Grade IV hematology.
* Hypersensitivity to any component of the formulation of study drug
* Prior history of taking any ARV for more than 10 days
* Concomitant administration of tenofovir (TDF).
* Refer to Section 6.4.1 which details all prohibited therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- Local Institution, Tallinn, Estonia
- France (4):
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Orléans
  - Local Institution, Paris
  - Local Institution, Suresnes
- Germany (4):
  - Local Institution, Düsseldorf
  - Local Institution, Hanover
  - Local Institution, Stuttgart
  - Local Institution, Ulm
- Local Institution, Dublin, Dublin, Ireland
- Italy (4):
  - Local Institution, Brescia
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
- Local Institution, Riga, Latvia
- Portugal (2):
  - Local Institution, Cascais
  - Local Institution, Porto
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- Spain (4):
  - Local Institution, Elche, Alicante
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
- United Kingdom (3):
  - Local Institution, Bristol, Avon
  - Local Institution, Edinburgh, Central
  - Local Institution, London, Greater London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 288 subjects were enrolled, of which 36 did not start Induction Phase Therapy (22 did not meet study criteria, 6 withdrew consent, 4 lost to follow-up, 3 had missing information, and 1 for investigator's decision).
Groups:
- Induction Treatment: Atazanavir (ATV) 300 mg + ritonavir (RTV) 100 mg, given once daily (QD) + 2 nucleoside reverse transcriptase inhibitors (NRTIs) during a 26- to 30-week Induction Phase
- Maintenance Treatment: Switch Regimen: Participants with confirmed undetectable viral load (ie, HIV-1 RNA viral load < 50 c/mL on 2 consecutive on-treatment measurements performed from Week 16 up until Week 28 of the Induction Phase), at the end of Induction Phase, who were then randomized to ATV 400 mg QD for an additional 48 weeks (continued previous NRTI).
- Maintenance Treatment: Continuation Regimen: Participants with confirmed undetectable viral load (ie, HIV-1 RNA viral load < 50 c/mL on 2 consecutive on-treatment measurements performed from Week 16 up until Week 28 of the Induction Phase) at the end of Induction Phase, who were then randomized to ATV 300 mg + RTV 100 mg QD for an additional 48 weeks (continued previous NRTI).
- Rescue Treatment: Participants without confirmed undetectable viral load at the end of Induction Phase were not randomized, but were offered to continue on ATV 300 mg + RTV 100 mg QD + 2 NRTIs for an additional 48 weeks (continued previous NRTI).
Period: Induction Phase
Arm/Group | Induction Treatment | Maintenance Treatment: Switch Regimen | Maintenance Treatment: Continuation Regimen | Rescue Treatment
Started | 252 | 0 | 0 | 0
Completed | 222 (Subjects randomized into Maintenance Phase=172 (87 ATV +85 ATV/RTV); Rescue Phase subjects=50) | 0 | 0 | 0
Not Completed | 30 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Poor/noncompliance | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Subject no longer meets study criteria | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Incarceration | 1 | 0 | 0 | 0
Not completed — Missing lab data | 1 | 0 | 0 | 0
Period: Maintenance Phase/Rescue Phase
Arm/Group | Induction Treatment | Maintenance Treatment: Switch Regimen | Maintenance Treatment: Continuation Regimen | Rescue Treatment
Started | 0 | 87 | 85 | 50
Completed | 0 | 78 | 72 | 41
Not Completed | 0 | 9 | 13 | 9
Not completed — Adverse Event | 0 | 1 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — RTV intake impossible | 0 | 0 | 1 | 0
Not completed — Poor/noncompliance | 0 | 3 | 2 | 3
Not completed — Pregnancy | 0 | 2 | 2 | 0
Not completed — Subject no longer meets study criteria | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Randomized Subjects: Switch Regimen: ATV 400 mg QD + 2 NRTIs
- Randomized Subjects: Continuation Regimen: ATV 300 mg + RTV 100 mg QD + 2 NRTIs
- Nonrandomized Subjects: All participants entering Rescue Phase after Induction Phase or discontinued during Induction Phase: ATV 300 mg + RTV 100 mg QD + 2 NRTIs
- Total: Total of all reporting groups
Arm/Group | Randomized Subjects: Switch Regimen | Randomized Subjects: Continuation Regimen | Nonrandomized Subjects | Total
Number analyzed (Participants) | 87 | 85 | 80 | 252
Age, Customized [Median (Full Range); unit: years] | 35 [21 to 66] | 35 [19 to 70] | 36 [20 to 71] | 36 [19 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 16 | 62
  Male | 65 | 61 | 64 | 190
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 73 | 70 | 66 | 209
  Black | 14 | 14 | 11 | 39
  Other | 0 | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Europe | 68 | 68 | 60 | 196
  Russian Federation | 19 | 17 | 20 | 56
Hepatitis B or C [Number; unit: Participants]
  Hepatitis B/C positive | 16 | 20 | 23 | 59
  Hepatitis B/C negative | 71 | 65 | 57 | 193
Baseline CD4 [Median (Full Range); unit: cells/mm3] | 255 [50 to 660] | 265 [64 to 490] | 227 [2 to 876] | 245 [2 to 876]
Baseline HIV-1 RNA [Median (Full Range); unit: log10c/mL] | 4.85 [3.51 to 5.88] | 4.86 [3.58 to 5.88] | 5.46 [3.74 to 5.88] | 4.95 [3.51 to 5.88]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL (c/mL) Through Week 48 of the Maintenance Phase
Description: Participants were considered successes unless they experienced treatment failure, or had missing Week 48 HIV-1 RNA. Treatment failure: virologic rebound (ie, 2 consecutive on-treatment HIV-1 RNA ≥ 50 c/mL, or last HIV-1 RNA ≥ 50 c/mL followed by discontinuation), or discontinuation before Week 48. Denominator included all randomized participants.
Time Frame: From the end of Induction Phase (Week 26 to Week 30 of Induction Phase treatment) through Week 48 of Maintenance Phase
Population: As-randomized population (as-randomized refers to the treatment regimen assigned at randomization).
Measure: Number; unit: Percentage of participants
Groups:
- Switch Regimen: ATV 400 mg QD + 2 NRTIs
- Continuation Regimen: ATV 300 mg + RTV 100 mg QD + 2 NRTIs
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 87 | 85
Percentage of participants | 78 | 75
Statistical Analysis 1: Comparison: Switch Regimen vs Continuation Regimen; The planned sample size of 178 randomized subjects (89 on each regimen) provides at least 80% power to demonstrate that the response rate on ATV is within a 15% margin of the response rate on ATV/RTV assuming: a 2-sided 95% confidence interval for the difference in response rate between treatment regimens (switch-continuation); a response rate of 85% in both the Continuation and Switch regimens; a margin of -15% for the difference in response rates between treatment regimens; Test type: Non-Inferiority or Equivalence — Efficacy at Week 48 on the Switch Arm was considered to be non-inferior to the Continuation Arm if the lower limit of the 95% Confidence Interval was greater than -15%; Normal approximation; Difference in proportions = 2.9, 95% CI [-9.8 to 15.5]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 c/mL Through Week 48 of the Maintenance Phase
Description: Participants were considered successes unless they experienced treatment failure, or had missing Week 48 HIV-1 RNA. Treatment failure: virologic rebound (ie, 2 consecutive on-treatment HIV-1 RNA ≥ 400 c/mL, or last HIV-1 RNA ≥ 400 c/mL followed by discontinuation), or discontinuation before Week 48. Denominator included all randomized participants.
Time Frame: From the end of Induction Phase (Week 26 to Week 30 of Induction Phase treatment) through Week 48 of Maintenance Phase
Population: As-randomized population. (As-randomized refers to the treatment regimen assigned at randomization.)
Measure: Number; unit: Percentage of participants
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 87 | 85
Percentage of participants | 86 | 81
Statistical Analysis 1: Comparison: Switch Regimen vs Continuation Regimen; Test type: Superiority or Other; Normal Approximation; Difference in Proportions = 5.0, 95% CI [-6.0 to 16.1]

3. Secondary Outcome: Kaplan-Meier Cumulative Proportion for Treatment Failure (HIV-1 RNA ≥50 c/mL) at Different Time Points Through Week 48 of the Maintenance Phase
Description: Treatment failure based on HIV-1 RNA ≥ 50 c/mL was defined as virologic rebound on or before Week 48 or discontinuation of study therapy before Week 48 for any reason. Time to treatment failure was analyzed using life tables. Measured Values shows the Kaplan-Meier cumulative proportion of participants without treatment failure up to the end of the respective interval.
Time Frame: Weeks 6-8, Weeks 14-16, Weeks 22-24, Weeks 30-32, Weeks 38-40, Weeks 46-48
Population: As-randomized population (as-randomized refers to the treatment regimen assigned at randomization).
Measure: Number; unit: Proportion of participants
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 87 | 85
Proportion of participants
  Proportion by Week 6-8 | 0.9655 | 0.9412
  Proportion by Week 14-16 | 0.9655 | 0.9176
  Proportion by Week 22-24 | 0.9540 | 0.9059
  Proportion by Week 30-32 | 0.9310 | 0.8824
  Proportion by Week 38-40 | 0.8506 | 0.8343
  Proportion by Week 46-48 | 0.8273 | 0.8176
Statistical Analysis 1: Comparison: Switch Regimen vs Continuation Regimen; Covariate in the model: treatment regimen; Test type: Superiority or Other; Cox Proportional Hazards Model; Cox Proportional Hazard = 0.97, 95% CI [0.50 to 1.88]

4. Secondary Outcome: Kaplan-Meier Cumulative Proportion for Treatment Failure (HIV-1 RNA ≥400 c/mL) at Different Time Points Through Week 48 of the Maintenance Phase
Description: Treatment failure based on HIV-1 RNA ≥ 400 c/mL was defined as virologic rebound on or before Week 48 or discontinuation of study therapy before Week 48 for any reason. Time to treatment failure was analyzed using life tables. Measured Values shows the Kaplan-Meier cumulative proportion of participants without treatment failure up to the end of the respective interval.
Time Frame: Weeks 6-8, Weeks 14-16, Weeks 22-24, Weeks 30-32, Weeks 38-40, Weeks 46-48
Population: As-randomized population. (As-randomized refers to the treatment regimen assigned at randomization.)
Measure: Number; unit: Proportion of participants
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 87 | 85
Proportion of participants
  Proportion by Week 6-8 | 0.9412 | 0.9885
  Proportion by Week 14-16 | 0.9176 | 0.9885
  Proportion by Week 22-24 | 0.9059 | 0.9770
  Proportion by Week 30-32 | 0.8824 | 0.9540
  Proportion by Week 38-40 | 0.8585 | 0.8966
  Proportion by Week 46-48 | 0.8585 | 0.8823
Statistical Analysis 1: Comparison: Switch Regimen vs Continuation Regimen; Covariate in the model: treatment regimen; Test type: Superiority or Other; Cox Proportional Hazards Model; Cox Proportional Hazard = 0.84, 95% CI [0.37 to 1.90]

5. Secondary Outcome: Change From End of Induction Phase in CD4 Cell Count at Week 48 of Maintenance Phase
Description: Change in CD4 Cell Count From End of Induction Phase at Week 48 of Maintenance Phase. Change=Week 48 maintenance Phase value - end of Induction Phase value; a decrease signifies worsening.
Time Frame: End of Induction Phase (Week 26 to Week 30 of Induction Phase treatment), Week 48 of Maintenance Phase
Population: As-randomized population (as-randomized refers to the treatment regimen assigned at randomization). Analysis uses observed values (participants included are those with CD4 measurements at end of Induction Phase and at Week 48 of Maintenance Phase).
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 76 | 68
cells/mm3 | 100 (14.7) | 92 (18.1)
Statistical Analysis 1: Comparison: Switch Regimen vs Continuation Regimen; Test type: Superiority or Other; Normal approximation; Difference in means at Week 48 = 7, 95% CI [-38 to 53]

6. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24 of Induction Phase
Description: Change From Baseline in CD4 Count at Week 24 of Induction Phase. Change=Week 24 Induction Phase value - Baseline value; a decrease signifies worsening.
Time Frame: Baseline, Week 24 of Induction Phase
Population: Analyses use observed values (participants included are those with CD4 measurements at Baseline and at the end of Induction Phase).
Measure: Mean (Standard Error); unit: cells/mm3
Groups:
- Randomized Subjects: All participants who were randomized at the end of Induction Phase to receive either Switch Regimen (ATV 400 mg QD + 2 NRTIs) or Continuation Regimen (ATV 300 mg + RTV 100 mg QD + 2 NRTIs)
- Nonrandomized Subjects: All participants entering Rescue Phase after Induction Phase or discontinued during Induction Phase (ATV 300 mg + RTV 100 mg QD + 2 NRTIs)
- Total: All participants treated with Induction Phase therapy (ATV 300 mg + RTV 100 mg QD + 2 NRTIs)
Arm/Group | Randomized Subjects | Nonrandomized Subjects | Total
Number analyzed (Participants) | 155 | 49 | 204
cells/mm3 | 170 (10.0) | 201 (18.5) | 177 (8.8)

7. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48 of Rescue Phase
Description: Change From Baseline in CD4 Count at Week 48 of Rescue Phase. Change=Week 48 Rescue Phase value - Baseline value; a decrease signifies worsening.
Time Frame: Baseline, Week 48 of Rescue Phase
Population: Analyses use observed values (participants included are those with CD4 measurements at Baseline and Week 48 of Rescue Phase).
Measure: Mean (Standard Error); unit: cells/mm3
Groups:
- Rescue Treatment: Nonrandomized participants completing Induction Phase (ATV 300 mg + RTV 100 mg QD + 2 NRTIs)
Arm/Group | Rescue Treatment
Number analyzed (Participants) | 38
cells/mm3 | 313 (26.6)

8. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 24 of the Induction Phase
Description: Change From Baseline in HIV-1 RNA at Week 24 of the Induction Phase. Change=Week 24 Induction Phase value - Baseline value; a decrease signifies improvement.
Time Frame: Baseline, Week 24 of Induction Phase
Population: Analyses use observed values (participants included are those with HIV-1 RNA measurements at baseline and at Week 24 of Induction Phase).
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | Randomized Subjects | Nonrandomized Subjects | Total
Number analyzed (Participants) | 151 | 47 | 198
log10 c/mL | -3.16 (0.046) | -3.35 (0.135) | -3.21 (0.048)

9. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 48 of the Rescue Phase
Description: Change From Baseline in HIV-1 RNA at Week 48 of the Rescue Phase. Change=Week 48 Rescue Phase value - Baseline value; a decrease signifies improvement.
Time Frame: \Baseline, Week 48 of Rescue Phase
Population: Analyses use observed values (participants included are those with HIV-1 RNA measurements at baseline and at Week 48 of Rescue Phase)
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | Rescue Treatment
Number analyzed (Participants) | 41
log10 c/mL | -3.71 (0.078)

10. Secondary Outcome: Treatment Outcomes Based on Viral Loads (HIV-1 RNA ≥50 c/mL) Through the End of Rescue Phase
Description: Treatment outcome is based on the first reason of failure. These analyses were performed using HIV-1 RNA of 50 c/mL to define suppression and virologic rebound.
Time Frame: Through Week 48 of Rescue Phase. Measurements were included from the end of Induction Phase through the last dose of Rescue Phase study therapy plus 4 days.
Measure: Number; unit: Participants
Arm/Group | Rescue Treatment
Number analyzed (Participants) | 50
Participants
  Suppression Maintained Through Week 48 | 29
  Suppression, then Virologic Rebound at/before Wk48 | 7
  Discontinuation Before Week 48 | 8
  Viral Suppression Never Achieved | 6

11. Secondary Outcome: Treatment Outcomes Based on Viral Loads (HIV-1 RNA ≥400 c/mL) Through the End of Rescue Phase
Description: Treatment outcome is based on the first reason of failure. These analyses were performed using HIV-1 RNA of 400 c/mL to define suppression and virologic rebound.
Time Frame: Baseline, Week 48 of Rescue Phase
Measure: Number; unit: Participants
Arm/Group | Rescue Treatment
Number analyzed (Participants) | 50
Participants
  Suppression Maintained Through Week 48 | 39
  Suppression, then Virologic Rebound at/before Wk48 | 2
  Discontinuation Before Week 48 | 9
  Viral Suppression Never Achieved | 0

12. Secondary Outcome: Time to Suppression (Confirmed HIV-1 RNA < 50 c/mL) During Treatment Phase
Description: Description: Time to suppression was measured from the first dose of Induction Phase study therapy to the first of the 2 consecutive measurements < 50 c/mL. Time to suppression was analyzed using life tables. Measured Values show the Kaplan-Meier cumulative number of treated participants without suppression up to the end of the respective interval.
Time Frame: Week 16-18, Week 24-26, Week 38-40, Week 64-66
Measure: Number; unit: Participants
Groups:
- Randomized Subjects: All participants who were randomized at the end of Induction Phase to receive either Switch Regimen (ATV 400mg QD + 2NRTIs) or Continuation Regimen (ATV 300mg + RTV 100mg QD + 2NRTIs)
- Nonrandomized Subjects: All participants entering Rescue Phase after Induction Phase or discontinued during Induction Phase (ATV 300mg + RTV 100mg QD + 2NRTIs)
Arm/Group | Randomized Subjects | Nonrandomized Subjects
Number analyzed (Participants) | 172 | 80
Participants
  Number of Participants Suppressed by Wk 16-18 | 131 | 3
  Number of Participants Suppressed by Wk 24-26 | 171 | 5
  Number of Participants Suppressed by Wk 38-40 | 172 | 31
  Number of Participants Suppressed by Wk 64-66 | 172 | 42

13. Secondary Outcome: Time to Suppression (Confirmed HIV-1 RNA < 400 c/mL) During Treatment Phase
Description: Time to suppression was measured from the first dose of Induction Phase study therapy to the first of the 2 consecutive measurements <400 c/mL. Time to suppression was analyzed using life tables. Measured Values show the Kaplan-Meier cumulative number of treated participants without suppression up to the end of the respective interval.
Time Frame: Week 16-18, Week 24-26, Week 30-32
Measure: Number; unit: Participants
Arm/Group | Randomized Subjects | Nonrandomized Subjects
Number analyzed (Participants) | 172 | 80
Participants
  Number of Participants Suppressed by Week 16-18 | 168 | 39
  Number of Participants Suppressed by Wk 24-26 | 171 | 54
  Number of Participants Suppressed by Wk 30-32 | 172 | 55

14. Secondary Outcome: Summary of Adverse Events During Induction Phase
Description: Summary of Adverse Events (AEs), Deaths, Serious AEs (SAEs), and AEs leading to study discontinuation. An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Measurements are included through the earlier of the last dose of Induction Phase study therapy plus 30 days or the first dose of Maintenance/Rescue Phase therapy (ie, up until 26 to 31 weeks + 30 days).
Population: Participants who received at least 1 dose of Induction Phase study therapy.
Measure: Number; unit: Participants
Arm/Group | Randomized Subjects | Nonrandomized Subjects | Total
Number analyzed (Participants) | 172 | 80 | 252
Participants
  Deaths | 0 | 3 | 3
  SAEs | 7 | 9 | 16
  SAEs related to study therapy | 0 | 2 | 2
  AEs leading to discontinuation | 0 | 9 | 9

15. Secondary Outcome: Summary of Adverse Events During Maintenance Phase
Description: as for outcome 14
Time Frame: Measurements are included from the end of Induction Phase (26 to 30 weeks after first dose) through the last dose of Maintenance Phase study therapy plus 30 days.
Population: Participants who received at least 1 dose of Maintenance Phase study therapy. As-treated population (as-treated refers to the actual treatment received during the Maintenance Phase).
Measure: Number; unit: Participants
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 87 | 85
Participants
  Deaths | 0 | 0
  Serious Adverse Events (SAEs) | 4 | 3
  SAEs related to study therapy | 0 | 0
  AEs leading to discontinuation | 1 | 4

16. Secondary Outcome: Summary of Adverse Events During Rescue Phase
Description: as for outcome 14
Time Frame: Measurements are included from the end of Induction Phase (26 to 30 weeks after the first dose therapy) through the last dose of Rescue Phase study therapy plus 30 days.
Population: Participants who received at least 1 dose of Rescue Phase study therapy
Measure: Number; unit: Participants
Arm/Group | Rescue Treatment
Number analyzed (Participants) | 50
Participants
  Deaths | 1
  SAEs | 2
  SAEs related to study therapy | 0
  AEs leading to discontinuation | 1

17. Secondary Outcome: Percent Change From End of Induction Phase in Fasting Lipids at Week 48 of Maintenance Phase
Description: Percent change in fasting lipids from end of Induction Phase to Week 48 of Maintenance Phase.Percent changes were calculated on the log scale and then back transformed to the original scale.Change=Week 48 maintenance Phase value - end of Induction Phase value; a decrease signifies worsening for HDL cholesterol and improvement for all other lipds.
Time Frame: Measurements were included from the end of Induction Phase (Week 26 to Week 30 of Induction therapy) through Week 48 of Maintenance Phase.
Population: Participants who received at least 1 dose of Maintenance Phase study therapy. As-treated population (as-treated refers to the actual treatment received during the Maintenance Phase). Analysis used last observation carried forward (LOCF) to replace missing values.
Measure: Mean (95% Confidence Interval); unit: percent change
Groups:
- Switch Regimen: ATV 400mg QD + 2NRTIs
- Continuation Regimen: ATV 300mg + RTV 100mg QD + 2NRTIs
Arm/Group | Switch Regimen | Continuation Regimen
Number analyzed (Participants) | 81 | 77
percent change
  Total Cholesterol | -4.7 [-8.28 to -1.02] | 1.4 [-1.88 to 4.78]
  HDL Cholesterol | 3.7 [-0.86 to 8.42] | 0.8 [-4.24 to 6.12]
  LDL Cholesterol | -0.7 [-6.7 to 5.8] | -2.1 [-7.10 to 3.26]
  Triglycerides | -27.0 [-33.21 to -20.19] | 9.8 [-1.35 to 22.23]
  Non-HDL Cholesterol | -7.4 [-12.15 to -2.48] | 1.1 [-3.34 to 5.65]

ADVERSE EVENTS:
Groups:
- Non-Randomized Participants: All participants entering Rescue Phase after Induction Phase or discontinued during Induction Phase (ATV 300mg + RTV 100mg QD + 2NRTIs)
Arm/Group | Switch Regimen | Continuation Regimen | Non-Randomized Participants
Serious Adverse Events (participants affected / at risk) | 7/87 | 5/85 | 11/80
Other Adverse Events (participants affected / at risk) | 72/87 | 75/85 | 52/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Switch Regimen (N=87) | Continuation Regimen (N=85) | Non-Randomized Participants (N=80)
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
DRUG DEPENDENCE (Psychiatric disorders) | 1 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
DUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 2
PNEUMONIA (Infections and infestations) | 1 | 1 | 2
MENINGITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
APPENDICEAL ABSCESS (Infections and infestations) | 0 | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Switch Regimen (N=87) | Continuation Regimen (N=85) | Non-Randomized Participants (N=80)
OCULAR ICTERUS (Eye disorders) | 15 | 18 | 6
BLOOD BILIRUBIN INCREASED (Investigations) | 32 | 33 | 17
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 | 8 | 7
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 | 3 | 7
DEPRESSION (Psychiatric disorders) | 5 | 2 | 3
JAUNDICE (Hepatobiliary disorders) | 4 | 9 | 3
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 5 | 5 | 5
HEADACHE (Nervous system disorders) | 11 | 13 | 8
NAUSEA (Gastrointestinal disorders) | 10 | 13 | 12
VOMITING (Gastrointestinal disorders) | 2 | 5 | 5
DIARRHOEA (Gastrointestinal disorders) | 14 | 14 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 9 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 5 | 4
SINUSITIS (Infections and infestations) | 2 | 5 | 0
BRONCHITIS (Infections and infestations) | 8 | 7 | 2
PHARYNGITIS (Infections and infestations) | 6 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 5 | 7 | 7
VIRAL INFECTION (Infections and infestations) | 3 | 2 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 4
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 4
RASH (Skin and subcutaneous tissue disorders) | 3 | 7 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 5
PYREXIA (General disorders) | 5 | 5 | 1
ASTHENIA (General disorders) | 7 | 10 | 8
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.